CLINICAL TRIAL: NCT03954262
Title: Evaluation of Autonomic Modulation After Propofol Induction Anesthesia With Target Controlled Infusion and Manually Bolus
Brief Title: Autonomic Modulation After Propofol Target Controlled Infusion and Bolus Administration
Status: Completed | Type: Observational
Sponsor: National Central University (Other)
Responsible Party: Principal Investigator, Hsin-Yi Wang, Taipei Veterans General Hospital, Principal Investigator, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2019-03-003CC
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia; Autonomic Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCI group: Group I received TCI at 5-6 ug/ml target effect concentration (Ce)
  Interventions: Behavioral: observation of propofol ANS response
- bolus group: groups II received an induction bolus of propofol (2-2.5mg/kg).
  Interventions: Behavioral: observation of propofol ANS response

INTERVENTIONS:
Behavioral: observation of propofol ANS response — received an induction bolus or TCI infusion of propofol

SUMMARY:
Some studies have compared the clinical profile during propofol induction anesthesia with Target-controlled infusion (TCI) and manually bolus showed similar control of anesthesia, such as depth of anaesthesia and hemodynamic stability, but did not use an objective measure of instantaneous autonomic activity during the brief time of induction anesthesia. In this study, TCI and manually bolus of propofol injection techniques during induction were studied with wavelet-based spectral analysis and the amplitudes of the pulse plethysmographic. The investigators hypothesized that during propofol induction anesthesia, the instantaneous ANS activities was more stable with TCI than traditional manually bolus

DETAILED DESCRIPTION:
Propofol induction anesthesia has been reported to be associated with cardiovascular depression and autonomic nervous system (ANS), which is an important neural control system for maintaining cardiovascular stability and plays a major role in regulating cardiovascular homeostasis. There are many methods for the administration induction of propofol, such as a manually bolus or target-controlled infusion (TCI) techniques. TCI devices could rapidly achieve and maintain the desired predicted concentration and is a more satisfactory technique to reduce the incidence of side effects and with the advantage of better hemodynamic control. More precise knowledge of how anesthetic agents modify ANS activity is important for understanding subsequent cardiovascular responses. However, there was no study using validated measurement of ANS index comparing propofol induction anaesthesia with TCI or manually bolus would have different effects on ANS.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgery under general anesthesia

Exclusion Criteria:

* recent administration of sedative or opioid drugs
* emergency surgery
* impairment of renal, hepatic, cardiac or respiratory function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects were selected from patients scheduled for surgery under general anesthesia. Exclusion criteria were recent administration of sedative or opioid drugs, emergency surgery and impairment of renal, hepatic, cardiac or respiratory function. No sedative or opioid drugs were administered before induction of anaesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of autonomic index with propofol induction-related sympathetic and parasympathetic imbalance- Assessed by continuous wavelet transform | about 5 minutes
  The presented work is aimed at applying instantaneous measures of heart rate variability data, as determined from the frequency domain analysis of the wavelet transform, to provide able to track fast autonomic effects during propofol induction.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei, R.o.c
  - Taipei Veterans General Hospital, Taiwan, Taipei